CLINICAL TRIAL: NCT02899949
Title: Real-world Data on Dapagliflozin: Characteristics and Health Outcomes of Patients With Type 2 Diabetes Treated With Dapagliflozin in Conjunction With Insulin
Brief Title: Health Outcomes of Patients With Type 2 Diabetes Treated With Dapagliflozin in Conjunction With Insulin
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Stewart Harris, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: ESR-15-11696
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: dapagliflozin; type 2 diabetes; real-world data
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Real-world data can supplement the knowledge gained from traditional randomized controlled trials. To date, only a couple of studies (Andrew et al. 2014 and Wilding et al. 2015) have been conducted assessing the use of dapagliflozin in the real-world clinical settings in the United Kingdom and no research has been done on the use of dapagliflozin in Canadian clinical practice settings.

To the investigators' knowledge, no real-world study exits assessing the impact of using dapagliflozin in conjunction with insulin in people with type 2 diabetes mellitus on dosage and frequency of insulin, oral antiglycemic agents and hypertension drugs. This study will use an electronic medical record-based data that contains demographic, drug coverage, vitals, lab results, medical problems and diabetes-related complications, and medication prescription information of patients with diabetes received care from all outpatient diabetes clinics in London Ontario, Canada to assess the impact of using dapagliflozin in conjunction with insulin in patients with type 2 diabetes mellitus on health outcomes, and medications dosing and frequency.

DETAILED DESCRIPTION:
Adult individuals (age≥18) with type 2 diabetes mellitus receiving care at the diabetes outpatient clinics at St. Joseph's Health Centre London (Canada) who have been treated with dapagliflozin in conjunction with insulin therapy will be selected from the Web DR researchable database for this study. Web DR is a diabetes-specific, web-based, researchable, electronic medical record and database. With no existing electronic medical record tailored for diabetes patients, the system was designed and implemented by the Centre for Diabetes, Endocrinology and Metabolism of St. Joseph's Health Care London. The St. Joseph's Centre for Diabetes, Endocrinology and Metabolism is the primary regional center for diabetes and endocrine disease management in Southwestern Ontario. Web DR is an electronic medical record with clinician-friendly pick-lists to enable structured electronic medical record data collection at the point of care, and is currently being used by 14 Endocrinologists and three Family Physician Diabetologists in the outpatient diabetes clinics at St. Joseph's Health Care London, Canada.

The baseline period will be 6 months to allow for more complete observation of comorbidities and medication use patterns. HbA1c, lipid, blood pressure, weight and other clinical indicators measured during the baseline period (closest to the date of dapagliflozin prescription) and follow-up period (3 and 6 months after prescription of dapagliflozin) will be extracted from the database. The last clinical value within the follow-up period and ≥30 days after the start of the medication data will be selected as follow-up information.

The type of insulin used and dosages prescribed during the study follow-up period will be extracted from the database to examine the insulin dosage prescription pattern and understand the use of insulin with dapagliflozin and its impact on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus >18 years of age, diabetes patients on insulin who initiated dapagliflozin due to a need of tighter glycemic control

Exclusion Criteria:

* glomerular filtration rate (GFR)<60, pregnancy, type 1

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study will use data from an EMR-based (Web DR) researchable database, which has been used to study patient's socioeconomic characteristics, treatment patterns and health outcomes of patients with diabetes. The Web DR de-identified researchable database contains integrated demographic, clinical and laboratory test result data of patients who received care from outpatient diabetes clinics in London, Ontario. The database includes more than 16,000 patients and their clinic visit information since 2000. Adult individuals (age>=18) with type 2 diabetes registered in Web DR who have been treated with dapagliflozin in conjunction with insulin therapy will be selected for this study.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
change in HbA1c value | baseline and 6 months
  mean change in HbA1c value at 6 months from baseline

SECONDARY OUTCOMES:
change in weight (kg) | baseline and 6 months
  mean change in weight at 6 months from baseline will be assessed
change in blood pressure (systolic and diastolic) | baseline and 6 months
  mean change in blood pressure at 6 months from baseline will be assessed
change in glomerular filtration rate | baseline and 6 months
  mean change in glomerular filtration rate at 6 months from baseline will be assessed
change in Insulin dose | baseline and 6 months
  change in Insulin dose (units) at 6 months from baseline will be assessed
Evidence of diabetic ketoacidosis documented | within the first 6 months from baseline
  Number of evidence of diabetic ketoacidosis within the first 6 months from baseline will be assessed
Evidence of genital infections documented | within the first 6 months from baseline
  Evidence of genital infections within the first 6 months from baseline will be assessed
Evidence of hypoglycemia events documented | within the first 6 months from baseline
  Number of hypoglycemia events documented within the first 6 months will be assessed
Evidence of urinary tract infection (UTI) documented | within the first 6 months from baseline
  Evidence of urinary tract infection (UTI)s documented within the first 6 months will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Harris, MD,MPH,FCFP, Principal Investigator — Lawson Research and Western University

IPD SHARING:
Plan to Share IPD: No